CLINICAL TRIAL: NCT01692678
Title: Multicenter, Open-label Study of YONDELIS (Trabectedin) in Subjects With Locally Advanced or Metastatic Liposarcoma or Leiomyosarcoma
Brief Title: A Study of Trabectedin (YONDELIS) in Patients With Locally Advanced or Metastatic Liposarcoma or Leiomyosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017269; ET743SAR3006 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2012-08-06; First posted 2012-09-25 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Advanced or Metastatic Liposarcoma or Leiomyosarcoma
Keywords: Advanced or Metastatic liposarcoma or leiomyosarcoma; Sarcoma; L-sarcoma; Liposarcoma; Leiomyosarcoma; Trabectedin; Dacarbazine; Yondelis; Chinese patients; Overall survival; Pharmacokinetics
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma; Sarcoma | interventions — Trabectedin; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabectedin (Part 1 and Part 2) (Experimental): Trabectedin will be administered at a dose of 1.5, 1.2 or 1.0 mg/m2 as a 24-hour intravenous infusion on Day 1 of each 21-day treatment cycle (ie, each treatment cycle being at least 21 days apart).
  Interventions: Drug: Trabectedin
- Dacarbazine (Part 2) (Active Comparator): Dacarbazine will be administered at a dose of 1 g/m2 as a longer than 30-minute intravenous infusion on Day 1 of each 21-day treatment cycle (ie, each treatment cycle being at least 21 days apart).
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Trabectedin — Type=exact number, unit=mg/m2, number=1.5, 1.2 or 1.0, form=solution, route=intravenous infusion. Trabectedin will be administered on Day 1 of each 21-day treatment cycle.
  Other Names: YONDELIS
  Arms: Trabectedin (Part 1 and Part 2)
Drug: Dacarbazine — Type=exact number, unit=g/m2, number=1, form=solution, route=intravenous infusion. Dacarbazine will be administered on Day 1 of each 21-day treatment cycle.
  Arms: Dacarbazine (Part 2)

SUMMARY:
The purpose of this study is to find the optimal dose of trabectedin for Chinese patients with locally advanced or metastatic L-sarcoma (liposarcoma or leiomyosarcoma) who were previously treated (in any order) with at least an anthracycline and ifosfamide containing regimen, or an anthracycline containing regimen and 1 additional cytotoxic chemotherapy regimen (Part 1) and to evaluate whether the overall survival (OS) of the trabectedin group is superior to dacarbazine group (Part 2).

DETAILED DESCRIPTION:
The study is divided into 2 separate parts (ie, Part 1 and Part 2). Part 1 is a dose finding part (to find the optimal dose) of trabectedin for Chinese patients, and Part 2 is a multicenter, randomized (the study medication is assigned by chance), active-controlled (an active substance that is compared with the study medication to test whether the study medication has a real effect in clinical study), parallel-group (a study comparing the response in two or more groups of patients receiving different interventions), open-label (all people know the identity of the intervention) bridging part comparing the efficacy and safety of the optimal dose of trabectedin with dacarbazine in the same population as in Part 1. The study (in both Part 1 and Part 2) will consist of a screening phase, a treatment phase and a follow-up phase. Part 1: Optimal dose (ie, maximum tolerated dose [MTD]) is determined from the following 3 dose levels: Dose level 1 (1.5 mg/m2), Dose level 2 (1.2 mg/m2), and Dose level 3 (1.0 mg/m2)of trabectedin. Cohorts of 6 patients will be treated at each dose level. To determine MTD, dose limiting toxicity (DLT; any pre-defined adverse event that occurs during the first cycle ie, Cycle 1) will be determined. In the first cohort of 6 patients, (a) if DLT is less than or equal to 1 at a dose level, it is considered as MTD (b) if DLT is greater than 2, patients will be de-escalated to next dose level (c) if DLT is equal to 2, 3 more patients will be included at that dose level and if there will be no DLT in those 3 patients, that dose level is considered as MTD. Part 2: If the optimal dose found in Part 1 is 1.5 mg/m2, approximately 48 patients will be randomly assigned to either the trabectedin (approximately 32 patients) or dacarbazine (approximately 16 patients) treatment group in Part 2. If the optimal dose found in Part 1 is below 1.5 mg/m2, 123 patients will be randomly assigned to either the trabectedin (approximately 82 patients) or dacarbazine (approximately 41 patients) treatment group. Safety will be evaluated by assessing adverse events, clinical laboratory test, multiple gated acquisition scans, electrocardiograms, vital signs, and physical examination throughout the study up to 30 days after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, unresectable, locally advanced or metastatic liposarcoma or leiomyosarcoma
* Treated in any order with at least: an anthracycline and ifosfamide containing regimen, or an anthracycline containing regimen and 1 additional cytotoxic chemotherapy regimen
* Measurable disease at baseline in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate recovery from prior therapy; all side effects (except alopecia) have resolved to Grade 1 or less according to the National Cancer Institute
* Adequate organ function and hepatic function

Exclusion Criteria:

* Prior exposure to trabectedin (both Part 1 and Part 2) or dacarbazine (Only Part 2)
* Less than 3 weeks from last dose of systemic cytotoxic therapy, radiation therapy, or therapy with any investigational agent
* Other malignancy within past 3 years (exceptions: basal or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ, or Federation Internationale de Gynecologie et d'Obstetrique (FIGO) Stage 1 carcinoma of the cervix)
* Known central nervous system metastasis
* Active or symptomatic viral hepatitis or chronic liver disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Optimal dose level (Maximum tolerated dose [MTD]) of trabectidin | From the date of dosing until 21days after the date of last patient enrolled
  MTD (1.5, 1.2 or 1.0 mg/m2) is determined by assessing Dose Limiting Toxicity (DLT).
Part 1: Overall survival | From the date of dosing upto 18 months after the last patient enrollment or 30 days after the last dose of study medication has been administered, whichever will be later
  Patients will be monitored for survival status at least every 60 days for the first 2 years after the last dose of study drug and every 90 days thereafter.
Part 2: Overall survival | From the date of randomization until the required number of events has occurred (approximately 32 if 1.5mg/m2, or 82 with below 1.5mg/m2) as assessed approximately for 6 months after the last patient enrollment
  Patients will be monitored for survival status at least every 60 days for the first 2 years after the last dose of study drug and every 90 days thereafter.

SECONDARY OUTCOMES:
Part 1: Progression free survival (PFS) | From date of dosing until the date of first documented progression or date of death from any cause, whichever comes first, as assessed up to 18 months after the last patient enrollment
  PFS is defined as the time from dosing to the occurrence of disease progression or death, whichever occurs first.
Part 2: Progression free survival (PFS) | From the date of randomization till the first documented disease progression or death whichever comes first until the required number of events, estimate of 6 months after the last patient enrollment
  PFS is defined as the time from randomization to the occurrence of disease progression or death, whichever occurs first.
Part 1: Time-to-progression (TTP) | From date of dosing until the date of first documented progression or date of death from any cause, whichever comes first, as assessed up to 18 months after the last patient enrollment
  Time-to-progression (TTP) is defined as the time between dosing and disease progression.
Part 2: Time-to-progression (TTP) | From the date of randomization till the first documented disease progression or death whichever comes first until the required number of events, estimate of 6 months after the last patient enrollment
  Time-to-progression (TTP) is defined as the time between randomization and disease progression.
Part 1: Objective Response Rate (ORR) | From date of dosing until the date of best response, as assessed up to 18 months after the last patient enrollment
  Objective Response Rate (ORR) is defined as having complete response or partial response as best overall response based on reconciled radiographic disease assessment.
Part 2: Objective Response Rate (ORR) | From date of dosing until the date of best response, as assessed up to 6 months after the last patient enrollment
  Objective Response Rate (ORR) is defined as having complete response or partial response as best overall response based on reconciled radiographic disease assessment.
Part 1: Duration of response (DR) | From date of dosing until the date of first documented progression or date of death from any cause, whichever comes first, as assessed approximately up to 18 months after the last patient enrollment
  Duration of response (DR) is defined only for patients who have CR or PR as best overall response and is calculated from the date of the first documentation of response to the date of disease progression or death, whichever occurs first.
Part 2: Duration of response (DR) | From the date of randomization till the first documented disease progression or death whichever comes first, assessed approximately up to 6 months after the last patient enrollment
  Duration of response (DR) is defined only for patients who have CR or PR as best overall response and is calculated from the date of the first documentation of response to the date of disease progression or death, whichever occurs first.
Part 1: Observed maximum plasma concentration (Cmax) | Days 1, 2, 3, 4, 5, 8 of first 2 treatment cycles
  Pharmacokinetic parameter Cmax of trabectedin will be determined
Part 1: Area under the plasma concentration-time curve (AUC) | Days 1, 2, 3, 4, 5, 8 of first 2 treatment cycles
  Pharmacokinetic parameter AUC of trabectedin will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (2):
- China (2):
  - Beijing
  - Shanghai

REFERENCES:
- See also: Multicenter, Open-label Study of YONDELIS (Trabectedin) in Subjects With Locally Advanced or Metastatic Liposarcoma or Leiomyosarcoma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=2432&filename=CR017269_CSR.pdf